CLINICAL TRIAL: NCT04913623
Title: Correlation of Intramedullary Pressure and Systemic Inflammatory Parameters as a Risk Indicator for Intraoperative and Early Postoperative Complications in Cemented and Non-cemented Femoral Stem of the Hip Arthroplasty
Brief Title: Correlation of Intramedullary Pressure and Systemic Inflammatory Parameters in Cemented Femoral Stem
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Clinical Centre of Kosova (Other)
Responsible Party: Principal Investigator, Skender Ukaj, Specialist of Orthopaedics and Trauma, University Clinical Centre of Kosova
Other Study IDs: 03/2021
Record Dates: First submitted 2021-04-05; First posted 2021-06-04 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-05

CONDITIONS: Arthroplasty Complications
MeSH Terms: interventions — Arthroplasty, Replacement, Hip; Arthroplasty

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Evaluation of the level of histamine, C-reactive protein (CRP) and leukocytes formula, IL1b, TNF alpha, IL6 and the reflection of changes of these parameters in the intra-operative course of hip replacement.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Correlation of intramedullary pressure and systemic inflammatory parameters in cemented THA
  Interventions: Procedure: Hip Replacement
- Correlation of intramedullary pressure and systemic inflammatory parameters in non cemented THA
  Interventions: Procedure: Hip Replacement

INTERVENTIONS:
Procedure: Hip Replacement — The hip replacement surgery is when a damaged hip is replaced with artificial one
  Other Names: Hip replacement surgery; Arthroplasty

SUMMARY:
The cemented femoral stem have impact on increase on systemic parameters.

Evaluation of the level of histamine, C-reactive protein (CRP) and leukocytes formula, IL1b, TNF alpha, IL6 and the reflection of changes of these parameters in the intra-operative course of hip replacement.

DETAILED DESCRIPTION:
Implantation of total endoprosthesis is a very common surgical procedure and is performed with and without bone cement.

In most cases during cementation of the femoral component there are changes in blood pressure, SpO2, heartbeat and other vital parameters which can cause complications during surgery.

Comparing the system parameters between the two groups and deriving these results will help the medical staff to be more professionally prepared to resolve possible complications.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria were as follows:

* All patients willing to participate who underwent cemented and uncemented THA,
* With no limit on age

Exclusion Criteria:

The exclusion criteria were patients with:

* Periprosthetic fractures,
* Pathological fractures
* THA revision
* ASA IV

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients are from the waiting list for surgery. All are included in the study with their consent The femoral component cemented or non-cemented is realized based on bone quality, age and its testing during surgery.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-03-23 (Actual); Primary Completion 2021-05-23 (Actual); Study Completion 2021-06-23 (Estimated)

PRIMARY OUTCOMES:
Change of systemic parameters during and after hip replacement (Histamine) | The measurement of these laboratory parameters 5 minutes before and 10 minutes after surgical procedures will reflect the impact of cements in the eventual post-surgical complications, such are embolism and other complications.
  Analysis of the impact of cement in different laboratory parameters such as histamine
Change of systemic parameters during and after hip replacement (CRP) | The measurement of these laboratory parameters 5 minutes before and 10 minutes after surgical procedures will reflect the impact of cements in the eventual post-surgical complications, such are embolism and other complications.
  Analysis of the impact of cement in different laboratory parameters such as C-reactive protein (CRP)
Change of systemic parameters during and after hip replacement (Leukocytes formula) | The measurement of these laboratory parameters 5 minutes before and 10 minutes after surgical procedures will reflect the impact of cements in the eventual post-surgical complications, such are embolism and other complications.
  Analysis of the impact of cement in different laboratory parameters such as changes of leukocytes formula
Change of systemic parameters during and after hip replacement (IL1b) | The measurement of these laboratory parameters 5 minutes before and 10 minutes after surgical procedures will reflect the impact of cements in the eventual post-surgical complications, such are embolism and other complications.
  Analysis of the impact of cement in different laboratory parameters such as IL1b
Change of systemic parameters during and after hip replacement (TNF alpha) | The measurement of these laboratory parameters 5 minutes before and 10 minutes after surgical procedures will reflect the impact of cements in the eventual post-surgical complications, such are embolism and other complications.
  Analysis of the impact of cement in different laboratory parameters such are TNF alpha
Change of systemic parameters during and after hip replacement (IL6) | The measurement of these laboratory parameters 5 minutes before and 10 minutes after surgical procedures will reflect the impact of cements in the eventual post-surgical complications, such are embolism and other complications.
  Analysis of the impact of cement in different laboratory parameters such as IL6.

SECONDARY OUTCOMES:
Difference of arterial pressure | The changes will be measured 5 minutes before implantation and during first 10 minutes after implantation
  Difference of arterial pressure after implantation of femoral component
Difference of changes of Leukocyte formula | The blood will be taken from patience 1 hour before and Post Operative Day One
  Difference of changes of Leukocyte formula after implantation of femoral component
Difference of SpO2 | The changes will be measured 5 minutes before implantation and during first 10 minutes after implantation]
  Difference of SpO2 after implantation of femoral component The changes will be measured by the device monitor connected to patient

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinical Center of Kosovo, Pristina, Kosovo

IPD SHARING:
Plan to Share IPD: Undecided